CLINICAL TRIAL: NCT04777877
Title: Exploring the Feasibility and Acceptability of Pain Neuroscience Education Delivered With a Virtual Reality Headset to Outpatient Physical Therapy Patients Treated for Low Back Pain: a Pilot Multi-site Implementation Trial
Brief Title: PNE Delivered With a VR Headset in Outpatient LBP Patients
Status: Completed | Type: Observational
Sponsor: Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, David Saul Binder, Principle Investigator, Spaulding Rehabilitation Hospital
Other Study IDs: 2021P000203
Record Dates: First submitted 2021-02-22; First posted 2021-03-02 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Pain Neuroscience Education delivered via a Virtual Reality Headset — Pain educational videos (5) and guided imagery 360 degree nature videos (5)

SUMMARY:
The primary objective of this study is to explore the feasibility and acceptability of the delivery of educational content using a virtual reality headset in the setting of an outpatient physical therapy (PT) course of care for chronic low back pain. We aim to collect both qualitative and quantitative data regarding: 1) specifics of device use in the course of PT care 2) acceptability of both the content and delivery method from the therapist and subject perspective 3) subject attributes to characterize the study population and explore possible associations with content responses and 4) changes in pain knowledge from pre to post intervention. Information learned in this pilot study will assist us in 1) improving the content and delivery method of a chronic pain education program 2) implementing the program across the Spaulding rehabilitation network and 3) designing a more rigorous effectiveness trial.

DETAILED DESCRIPTION:
Study staff physical therapists will identify potential subjects upon completion of a standard physical therapy evaluation on patients referred for low back pain. Spaulding Outpatient sites in Malden, Quincy YMCA and Charlestown will participate.

* Inclusion criteria: 1) pain lasting > 3 months and 2) > 18 years of age
* Exclusion criteria: 1) inability to understand and communicate in English 2) inability to provide informed consent Individuals who meet the inclusion/exclusion criteria will receive an information study sheet, the full consent form for reference, and hear a brief explanation of the study from the treating study staff physical therapist. It will be emphasized that study participation is completely voluntary and refusal to participate will in no way impact their care at that clinic site or other MGB facilities either now or in the future.

SUBJECT ENROLLMENT

Once an eligible subject is identified, the evaluating study staff physical therapist will briefly introduce the study and provide the study information sheet and full consent form for review. Interested individuals will be contacted by phone by study staff. Study staff obtaining consent will discuss the details of the study with the individual using the full consent form and study information sheet as a guide and will cover all of the required elements of informed consent, including the purpose of the research, the study procedures, risks and benefits associated with participation, and answer study-related questions. Subjects will be advised that their clinical care will not be affected in any way if they decide to participate or decline participation, and that participation can be discontinued at any time. The principal investigator's and consenting study staff's contact information will be provided on the information sheet and consent form, and other study staff will provide their contact information as appropriate. The study will be explained in detail and the individual will be given the chance to ask any questions. Informed consent will be obtained verbally over the phone due to the minimal study risk, low study burden, and the necessity of limiting in-person contact. Study staff will document verbal consent by electronically signing a copy of the IRB approved telephone information consent document which will be electronically stored in a protected Dropbox file that only study staff will have access to. Paper consent forms will not be stored. A copy will be securely emailed via Outlook to the treating study staff physical therapist. This copy will be printed and provided to the subject in-person by the treating study staff physical therapist at the subject's next scheduled physical therapy visit.

Due to the minimal risk involved, informed consent may be given with less than 12 hours of notice, or they may be given additional time to consider.

STUDY PROCEDURES

Study staff physical therapists will be informed of enrollment. Once enrolled, subjects will complete the Keele STarT back questionnaire and a pain knowledge check. The pain education content will be delivered via the Oculus Go virtual reality (VR) headset at the beginning or end of the subjects scheduled PT appointments. There will be no added costs for content delivery and no additional study visits will be required outside of the regularly scheduled PT visits. Upon completing the pain education series, subjects will complete a feedback survey and a post-pain knowledge check. Study staff physical therapists will complete a survey for each enrolled subject.

Additionally, demographic information will be collected from the Epic electronic health record (EHR) such as: age, gender, educational level, relevant past medical history, results of relevant images, and pertinent physical therapy evaluation and treatment information that is standard of care for this patient population. This information will be used to characterize the study sample and begin to identify important attributes that may have more relevance regarding the response to the content.

ELIGIBILITY:
Inclusion Criteria:

* pain lasting > 3 months
* 18 years of age or older

Exclusion Criteria:

* inability to understand and communicate in English
* inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: chronic low back pain patients referred for outpatient physical therapy
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-02-18 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Pain knowledge and beliefs questionnaire | Through study completion; an average of 4 clinical sessions delivered over 2 to 4 weeks
  assesses change in subject's knowledge and beliefs about pain

CONTACTS AND LOCATIONS:
Overall Officials: David Binder, MD, Principal Investigator — Spaulding Rehabilitation Hospital
Locations (1):
- Spaulding Rehabilitation Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brown L, DiCenso-Fleming T, Ensign T, Boyd AJ, Monaghan G, Binder DS. Chronic pain education delivered with a virtual reality headset in outpatient physical therapy clinics: a multi-site exploratory trial. Am J Transl Res. 2023 May 15;15(5):3500-3510. eCollection 2023. PMID 37303618